CLINICAL TRIAL: NCT04833699
Title: The Effect of Hot Pack Application of Umbilical Region on Postoperative Ileus in Patients Undergoing Surgery for Gynecologic Malignancies: a Randomized Controlled Trial
Brief Title: The Effect of Hot Pack Application on Postoperative Ileus Undergoing Surgery for Gynecologic Malignancies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erzincan Military Hospital (Other)
Responsible Party: Principal Investigator, Kemal GUNGORDUK, KG, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MUGLA-3
Record Dates: First submitted 2021-03-27; First posted 2021-04-06 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Postoperative Ileus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Group A or the control group did not pick up any therapy except our clinical standard postoperative care (ERAS protocol)
- Study (Experimental): Group B served as the hot pack group boiled tap water (80 °C) was put in a rubber water bag with a fluffy cover (Fig. 1), and placed on the patient's abdomen at 3, 6, 9, and 12 h after the surgical procedure for 30 minutes in addition to clinical standard postoperative care (ERAS protocol).
  Interventions: Other: rubber water bag

INTERVENTIONS:
Other: rubber water bag — bboiled tap water (80 °C) was put in a rubber water bag with a fluffy cover (Fig. 1), and placed on the patient's abdomen at 3, 6, 9, and 12 h after the surgical procedure for 30 minutes in addition to clinical standard postoperative care (ERAS protocol)
  Arms: Study

SUMMARY:
Postoperative ileus (POI), is an extensively known complication characterized by an impairment of normal gastrointestinal motor activity after abdominal surgery and may also occur after surgery at other sites due to non-mechanical causes. [1]. This clinical asset has been linked to prominent perioperative morbidity with the following financial burden owing to extended hospitalization [1]. Furthermore, POI can postpone adjuvant treatments, such as chemotherapy in patients who went through surgery for cancers.

Abdominal tenderness and distension, nausea and vomiting, delay in the passage of flatus and stool, and intolerance to solid food are the prime symptoms of POI [1-3]. It is generally transient, but if prolonged, can cause surgical incision dehiscence, intestinal anastomotic fistula, abdominal cavity infection, intestinal ischemia, aspiration pneumonia, and other serious complications [4-6]. Hence, many clinicians have focused on averting POI. Many studies have analyzed preventive methods, such as preoperative mobilization of the patient, adequate pain control, gum chewing, epidural anesthesia, coffee consumption, and motility agents such as metoclopramide and alvimopan [7-15]. For all the manifold remedy approaches, POI maintains a difficult clinical challenge that compromises the rapid improvement of patients who underwent abdominal surgery.

Recently, thermal attempts have been employs for several situations such as inflammatory bowel disease, chronic pelvic pain, and abdominal pain [16]. It may be used in two different ways; whole body or local. Local thermal therapy can be carried out by hot pack or paraffin [17]. It has been demonstrated that local thermotherapy abate myotonia, enhances circulation, and eases pain by expediting the removal of the pain-producing substance. Local thermal therapy is widely used for a number of conditions such as pain, nausea, vomiting, and some bowel diseases in traditional Chinese medicine [18].

ELIGIBILITY:
Inclusion Criteria:

* patiens aith aged ≥18 years olds
* patients undergoing elective exhaustive staging surgery (total hysterectomy (Type A-C2), systematic pelvic para-aortic lymphadenectomy ± bilateral salpingo-oophorectomy and ± omentectomy by abdominal approach containing either open or laparoscopic surgery.

Exclusion Criteria:

* ASA score >3,
* chronic constipation (defined as ≤2 bowel movements per week),
* inflammatory bowel disease,
* irritable bowel syndrome,
* compromised liver function,
* clinically significant cardiac arrhythmia,
* Thyroid disorder,
* History of abdominal bowel surgery,
* previous abdominal irradiation,
* previous neoadjuvant chemotherapy or hyperthermic intraperitoneal chemotherapy,
* Performed upper abdominal surgery
* The covid-19 positive test result,
* bowel anastomosis.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
time to the first passage of flatus after surgery | up to 72 hours
  Patients were checked hourly for bowel sounds by auscultation and were asked to note the time of first flatus and defecation and to inform the clinical nurses or an assistant.

SECONDARY OUTCOMES:
The time to tolerate a solid diet | Up to 5 days
  The time to tolerate a solid diet was measured from the end of operation, referred to the time when the patient awoke from anesthesia, until the patient tolerated intake of solid food (any food that required chewing) without vomiting
The time to the first bowel movement | up to 72 hours
  The time to the first bowel movement was referred to the time to the first audible bowel sound during routine postoperative care. Patients were checked hourly for bowel sounds by auscultation and were asked to note the time of first flatus and defecation and to inform the clinical nurses or an assistant.

CONTACTS AND LOCATIONS:
Locations (1):
- Mugla Sıtkı Kocman University Education and Research Hospital, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gungorduk K, Selimoglu B, Gulseren V, Yasar E, Comba C, Ozdemir IA. Effect of abdominal hot pack application on gastrointestinal motility recovery after comprehensive gynecologic staging surgery. Int J Gynaecol Obstet. 2024 Mar;164(3):1108-1116. doi: 10.1002/ijgo.15181. Epub 2023 Oct 6. PMID 37800343